CLINICAL TRIAL: NCT06565143
Title: Effect of Transcranial Alternating Current Stimulation(tACS) for Early Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Director of medical psychological department, Anhui Medical University, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: AHMU-TACS-AD
Record Dates: First submitted 2024-08-14; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Transcranial Alternating Current Stimulation; Electroencephalography; Early Alzheimer's Disease
Keywords: Transcranial Alternating Current Stimulation; Electroencephalography; Neuropsychology; Early Alzheimer's Disease; Alzheimer's Disease Assessment Scale-Cognitive Subscale; Working Memory
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcranial alternating current stimulation-Real (Active Comparator): Participants will receive real tACS once daily for 14 days
  Interventions: Device: Transcranial alternating current stimulation
- transcranial alternating current stimulation-Sham (Sham Comparator): Participants will receive sham tACS once daily for 14 days
  Interventions: Device: Sham transcranial alternating current stimulation

INTERVENTIONS:
Device: Transcranial alternating current stimulation — Transcranial alternating current stimulation (tACS) is a non-invasive brain stimulation tool that alters cortical excitability and activity via application of weak alternating currents.
  Arms: transcranial alternating current stimulation-Real
Device: Sham transcranial alternating current stimulation — In the sham condition, tACS was delivered only during the ramp-up and ramp-down periods (30s); no current was delivered during the 30-minute intervention.
  Arms: transcranial alternating current stimulation-Sham

SUMMARY:
To investigate the clinical effect neural mechanism of transcranial alternating current stimulation in early Alzheimer's disease

DETAILED DESCRIPTION:
Upon meeting the inclusion criteria and providing informed consent, each participant will complete a series of cognitive assessments and tACS at the First Affiliated Hospital of Anhui medical university. Patients were randomly allocated to tACS group and the sham group. There are about 20 patients in each group. For the all patients, allocation was by coin toss. Patients were studied using a double-blind design. Study participants and all personnel responsible for the clinical care of the patient remained masked to allocated condition and allocation parameters. Only tACS administrators had access to the randomization list; they had minimal contact with the patients, and no role in cognitive and symptom assessments. Each patient would be treated for continuous 14 days by tACS.

Before the tACS treatment, a series of cognitive assessments and neuropsychological tests were obtained by a trained investigator to assess baseline. Each assessment will involve a set of assessment tools, the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) as the primary outcome measure and various other tasks and questionnaires to measure cognition (including MoCA,MMSE, DS, Stroop test, TMT, BNT-30, VFT, CDT,JLOT. Form H,HVOT), memory (CAVLT, LMT), emotion(HAMA-17,HAMD-14,GDS-30), behavioral and psychological symptoms(NPI), and treatment tolerability. All the tests are conducted in two days. The patient received resting EEG data collection. After the last treatment, the MoCA, and associative memory were obtained, as well as the Global Index of Safety to assess adverse events of the treatment. Patients were instructed to focus their answers on the past 14 days. The patients had also receiving a battery measure of neuropsychological tests, resting EEG. Two months after the last treatment, participants were interviewed to obtain the same assessment as before. They were instructed to focus their answers on the past months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject diagnosed with early Alzheimer's disease or related diseases according to NIA-AA criteria.
2. Subjects must have a MMSE score between 10 and 27,indicating mild cognitive impairment or dementia.
3. CDR score ≤ 2.
4. Subject under treatment by IAChE for at least 3 months.
5. psychotropic treatments are tolerated if they were administered and unchanged for at least 3 months.

Exclusion Criteria:

1. CDR > 2
2. Any history or clinical signs of other severe psychiatric illnesses (like major depression,psychosis or obsessive compulsive disorder).
3. History of head injury,stroke,or other neurologic disease.
4. Organic brain defects on T1 or T2 images.
5. History of seizures or unexplained loss of consciousness.
6. Implanted pacemaker,medication pump,vagal stimulator,deep brain stimulator.
7. Family history of medication refractory epilepsy.
8. History of substance abuse within the last 6 months.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Alzheimers Disease Assessment Scale Cognitive section(ADAS-Cog) | changes from baseline at 14 days and 12 weeks post-treatment
  The changes in Alzheimers Disease Assessment Scale Cognitive section (ADAS-Cog) will constitute the major research outcome measure used to assess response to transcranial alternating current stimulation (tACS).The ADAS-Cog scale is a scale used for clinical assessment of dementia patients with some memory efficiency tests, which can be used as an objective assessment of memory. The scale is considered a tool capable of providing a specific assessment of the severity of cognitive and non-cognitive behavioral impairments in people with Alzheimer's disease or dementia. The advantage of the ADAS-Cog compared to other scales used in the same clinical area is that its score quantifies clinical and impressionistic aspects of the patient assessed by the examiner, as well as objectively defined cognitive characteristics. The higher the ADAS-Cog score, the worse the cognitive function. The minimum value is 0 and the maximum is 86.

SECONDARY OUTCOMES:
electroencephalography | changes from baseline at 14 days and 12 weeks post-treatment
  EEG recordings were obtained from each subject based on 64 electrode locations of the International 10-20 system (sampling frequency 1000Hz).The recorded EEG data were filtered with a second order band-pass Butterworth filter with cutoff frequencies of 0.5 and 60 Hz. For each testing condition, data with muscular, ocular and other types of artifacts were manually discarded and 60 seconds of stationary EEG signal were selected. Only these segments were accepted for further analysis.
  The analysis in the frequency domain was performed using Welch's periodogram method. Recordings were segmented into tracts of 10 seconds each, windowed with a Hanning window, with 50% overlap. The relative powers of the spectral components in the typical spectral bands delta (δ: 0.5-4 Hz), theta (θ: 4-8 Hz), alpha1 (α1: 8-10.5 Hz), alpha2 (α2: 10.5-13 Hz), beta1 (β1: 13-20 Hz), beta2 (β2: 20-30 Hz) and gamma (γ: 30-60 Hz) were computed by dividing the absolute power in each band by the total power.
Associative Memory | changes from baseline at 14 days and 12 weeks post-treatment
  The associative memory test uses facial cue word recall. The subjects memorized 20 photos of faces displayed on a screen in gray scale for 4 seconds each. When each card was presented, a common word appeared alongside the face. The subjects had to remember associations between faces and words by association. After a delay of about a minute after the study ended, the subjects were shown 12 of the same faces in different random orders, instructing them to recall the words that appeared with each face during the study. Recorded the correct number of words each face recalled. The faces were taken from a database of 24 amateur models. Each test format included only male or female faces.
MMSE(Mini Mental State Examination) | changes from baseline at 14 days and 12 weeks post-treatment
  The full name of MMSE is mini-mental state examination, and the scale consists of 30 subject, include the following seven aspects: time orientation, place orientation,immediate memory,attention and calculation,delay memory,language, visual space.One point is awarded for each question correctly answered during MMSE evaluation. If subject give the wrong answer or don't know answe he/she awarded 0 score, scope of scale score of 0 to 30 points. The higher the score, the better.
LMT (Logic Memory Test) | changes from baseline at 14 days and 12 weeks post-treatment
  The changes in LMT will constitute the secondary research outcome
DST (Digital Span Test; Forward and Backward) | changes from baseline at 14 days and 12 weeks post-treatment
  The changes in DST will constitute the other research outcome.
TMT (Trail Making Test) | changes from baseline at 14 days and 12 weeks post-treatment
  The Trail Making Test (TMT) is divided into two parts, part A and part B. Part A requires the subject to connect 25 Numbers on the paper in sequence, and part B requires the subject to connect 25 Numbers of different colors alternately in sequence. The time it takes for the subject to complete all the Numbers is the subject's final score.
HAMD (Hamilton Depression Scale) | changes from baseline at 14 days and 12 weeks post-treatment
  The changes in HAMD will constitute the other research outcome. The examination content consists of 17 questions (about 10 minutes), with a full score of 52. The higher the score, the more severe the depressive symptoms are.
HAMA (Hamilton Anxiety Scale) | changes from baseline at 14 days and 12 weeks post-treatment
  The changes in HAMD will constitute the other research outcome. The examination content consists of 14 questions (about 10 minutes), with a full score of 56. The higher the score, the more severe the anxiety symptoms are.
NPI (Neuropsychiatric Inventory) | changes from baseline at 14 days and 12 weeks post-treatment
  The changes in HAMD will constitute the other research outcome.
changes in Montreal Cognitive Assessment (MoCA) | changes from baseline at 14 days and 12 weeks post-treatment
  MoCA was developed by Nasreddine et al. based on clinical experience and reference to the MMSE cognitive items and scores, and the final version was finalized in November 2004. We adopted a localized version (Mandarin version，includes 2 alternative versions) in line with the Chinese cultural background.It includes 11 inspection items in 8 cognitive fields, including visual structure skills, executive function, naming, attention and calculation, language, abstract thinking, memory, and orientation. With a total score of 30 or more than 26, it is normal. Anyone who has been education for less than 12 years will need to add one point to his final score.
GDS(Geriatric depression scale) | changes from baseline at 14 days and 12 weeks post-treatment
  The Geriatric Depression Scale (GDS) was created in 1982 by Brank et al. and is dedicated to screening for depression in the elderly. The most suitable feelings for the elderly in the past week were evaluated.There are 30 items in the scale, the total score is 30 points. The higher the score, the more obvious the depressive symptoms. It is generally considered that less than 10 points is normal.
JLOT(Judgment of line Judgment of line orientation test orientation test) | changes from baseline at 14 days and 12 weeks post-treatment
  The JLOT test was determined by Benton et al. in 1994. There are two versions of H and V. The difference is that the order in which the pictures are presented is different. Each version contains 35 images, of which the official test consists of 30 images, and the other 5 images are for the participants to learn. The final score is the correct number of subjects to answer, the full score is 30 points, the higher the score, the better the space perception ability of the subject.
HVOT(Hooper visual organization test Hooper visual organization test) | changes from baseline at 14 days and 12 weeks post-treatment
  The changes in HVOT(Hooper visual organization test Hooper visual organization test) will constitute assess response to rTMS the secondary research outcome measure.HVOT is a cognitive test used to evaluate the perceived structure of the subject. It consists of 30 items，and each question is 1 point and the total score is 30 points. The final score is the correct number of subjects to answer, the full score is 30 points, the higher the score, the better the space perception ability of the subject.
The Stroop color test | changes from baseline at 14 days and 12 weeks post-treatment
  The Stroop color word test was developed by Stroop in 1935 and is used to evaluate the attention function of the subject. The subject is required to correctly read the target color on the stimulus card and record the completion time. The final completion time is the score of the participant. The shorter the time used, the better the performance of the subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China